CLINICAL TRIAL: NCT00879827
Title: Immunogenicity and Reactogenicity of GSK Biologicals' DTPa-HBV-IPV and Hib Vaccines When Administered Concomitantly to Healthy Infants Administered as a Three-dose Primary Vaccination Course at the Age of 1.5, 3.5 and 6 Months
Brief Title: Immunogenicity and Reactogenicity of GSK Bio DTPa-HBV-IPV and Hib Vaccines When Coadministered to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 217744/049
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Diphtheria; Poliomyelitis; Hepatitis B; Tetanus; Acellular Pertussis
MeSH Terms: conditions — Diphtheria; Poliomyelitis; Hepatitis B; Tetanus

ARMS (1):
- Single Group (Experimental)
  Interventions: Biological: Pediarix TM, Infanrix penta TM; Biological: Hiberix TM

INTERVENTIONS:
Biological: Pediarix TM, Infanrix penta TM — The vaccines were administered according to a 3-dose schedule at 1.5, 3.5 and 6 months of age.
Biological: Hiberix TM — The vaccines were administered according to a 3-dose schedule at 1.5, 3.5 and 6 months of age.

SUMMARY:
The purpose of this study is to evaluate the immune response and reactogenicity of GSK Biologicals' DTPa-HBV-IPV combined pentavalent vaccine and Hib tetanus conjugate vaccine, administered concomitantly as a three-dose primary vaccination course.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between 6 and 8 weeks of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the parents or guardians of the subject.
* Born after a normal gestation period (between 36 and 42 weeks).

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the first dose of study vaccine.
* Administration of chronic immunosuppressants or other immune-modifying drugs since birth or planned administration during the study.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of vaccine(s) and ending 30 days after.
* Previous vaccination against diphtheria, tetanus, pertussis, polio or Haemophilus influenzae type b.
* History of, or intercurrent, diphtheria, tetanus, pertussis, hepatitis B, polio and/or Haemophilus influenzae type b.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection.
* Major congenital defects
* Serious chronic illness
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Acute disease at the time of enrollment.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2000-09; Primary Completion 2001-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Anti-PT, anti-FHA and anti-PRN antibody titers. | One month after the 3rd dose of the primary vaccination course
Anti-diphtheria toxoid and anti-tetanus toxoid antibody titers | One month after the 3rd dose of the primary vaccination course
Anti-HBs antibody titers | One month after the 3rd dose of the primary vaccination course
Anti-polio virus types 1, 2 and 3 antibody titers | One month after the 3rd dose of the primary vaccination course
Anti-PRP antibody titers | One month after the 3rd dose of the primary vaccination course

SECONDARY OUTCOMES:
Occurrence of solicited adverse events | During the 4-day follow-up period after each dose
Occurrence of unsolicited adverse events | During the 30-day follow-up period after each dose
Occurrence of Serious Adverse Events | Over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Shao PL, Lu CY, Hsieh YC; Taiwan Infanrix-049 Study Group; Bock HL, Huang LM. Immunogenicity and reactogenicity of diphtheria-tetanus-acellular pertussis-hepatitis B-inactivated poliovirus and Haemophilus influenzae type B. J Formos Med Assoc. 2011 May;110(5):336-41. doi: 10.1016/S0929-6646(11)60050-8. PMID 21621155
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 217744/049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 217744/049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 217744/049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 217744/049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 217744/049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register